CLINICAL TRIAL: NCT00318838
Title: A Double-blind, Randomized, Parallel-group, Placebo-controlled, Multiple-dose Study to Assess the Effect of 125 mg/Day Orally Administered Azimilide Dihydrochloride on Renal Function and Hemodynamics in Healthy Volunteers
Brief Title: Effect of Azimilide Dihydrochloride on Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Jose Brum, MD, Procter and Gamble Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006022
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — azimilide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo tablet every 12 hours for 3 days followed by placebo tablet every 24 hours for three days
  Interventions: Drug: Placebo
- 2 (Experimental): 125 mg azimilide tablet every 12 hours for 3 days followed by 125 mg azimilide tablet every 24 hours for three days
  Interventions: Drug: Azimilide dihydrochloride

INTERVENTIONS:
Drug: Azimilide dihydrochloride — 125 mg azimilide tablet every 12 hours for 3 days followed by 125 mg azimilide tablet every 24 hours for three days
  Arms: 2
Drug: Placebo — Placebo tablet every 12 hours for 3 days followed by placebo tablet every 24 hours for three days
  Arms: 1

SUMMARY:
This study will assess the effect of multiple dosing of 125 mg azimilide on glomerular filtration rate (GFR) and total creatinine clearance (GFR + active secretion) in healthy subjects. Also, it will assess the effect of multiple dosing of 125 mg azimilide on renal hemodynamics (RPF) in healthy subjects.

DETAILED DESCRIPTION:
This is a double-blind, parallel-group, placebo-controlled, multiple-dose, single-site study in healthy male and female volunteers. Oral azimilide 125 mg or placebo will be administered every 12 hours for 3 days, followed by 125 mg every 24 hours for 3 days. The study will include a total of 21 healthy subjects (14 active and 7 placebo), all of whom will be confined at the study center for 9 nights.

ELIGIBILITY:
Inclusion Criteria:

* Male or hysterectomized or post-menopausal (last menstrual period > 1 year) female
* Between 18 and 45 years of age, inclusive, at screening
* In good general health based on medical history, physical examination and laboratory evaluation
* Body mass index between 18 and 32 (kg/m2), inclusive
* Willing and able to fulfill the requirements of the protocol and provide written consent

Exclusion Criteria:

* History of diabetes, cardiovascular, hepatic, renal, or gastrointestinal disease
* History of use of tobacco or nicotine-containing products within the past 3 months
* Alcohol or illicit drug abuse or a reported habitual alcohol intake greater than 1.5 oz. (ethanol equivalent) per day (e.g., 24 ozs. of beer, 10 ozs. of wine, or 3 ozs. of hard liquor) within the past 2 years.
* History of a clinically significant (in the opinion of the investigator) allergic reaction to any drug or multiple food/drug, contrast media agents, PAH, iodine or shell fish.
* Clinically significant abnormality upon physical examination that, in the investigator's opinion, would interfere with the conduct of the study
* Corrected QT-interval (QTc) > 440 msec (QT interval corrected for heart rate using Bazett's formula).
* Clinically significant abnormality on screening 12-lead electrocardiogram (ECG); presence of discernable U wave that (in the investigator's opinion) would interfere with accurate measurement of QT at baseline and/or after treatment.
* Personal or family history of long QT syndrome
* Absolute neutrophil count < 1500/mm3
* Potassium or magnesium value(s) outside the laboratory normal range
* Any other laboratory value(s) outside the laboratory normal range considered clinically significant by the investigator (serum chemistry, hematology, coagulation, or urinalysis.
* Serology positive for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) screen.
* If female, positive urine or serum pregnancy test
* Positive urine screen for drugs of abuse
* Reported use of any prescription drug or herbal preparations within 14 days prior to dosing or any non-prescription drug or vitamin within 7 days prior to dosing.
* Reported use of any known enzyme-inducer, enzyme-inhibitor, or other investigational drug within 30 days prior to dosing, or reported chronic exposure to enzyme-inducers such as paint solvents or pesticides within 30 days of dosing.
* Blood donation of approximately 400 mL or more within 4 weeks or plasma donation of 200 mL or more within 2 weeks prior to dosing.
* Acute illness within 2 weeks prior to dosing
* History or presence, upon clinical evaluation, of any illness that might impact the safety of test product administration or evaluability of drug effect based on the investigator's discretion.
* Has participated in another investigational drug study protocol within 30 days of admission.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To assess the effect of multiple dosing of 125 mg azimilide on glomerular filtration rate and total creatinine clearance in healthy subjects | 6 days

SECONDARY OUTCOMES:
To assess the effect of multiple dosing of 125 mg azimilide on renal hemodynamics in healthy subjects | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Brum, MD, Study Director — Procter and Gamble
Locations (1):
- Parexel CPRU, Harbor Hospital Center, Baltimore, Maryland, United States